CLINICAL TRIAL: NCT06577766
Title: A Randomised, Placebo Controlled, Double Blinded Study Assessing the Safety, Tolerability and Pharmacokinetics of Single and Multiple Subcutaneous Doses of NNC0638-0355 in Participants With Overweight or Obesity
Brief Title: A Research Study on How NNC0638-0355, a New Medicine, Works in People Living With Overweight or Obesity
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9638-7569; U1111-1296-8015 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-08-28; First posted 2024-08-29 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NNC0638-0355 (Experimental): Participants will be randomized to receive NNC0638-0355. The study will be conducted in 4 parts. Part A: Single ascending dose (SAD) Part B, C and D: Multiple ascending dose (MAD).
  Interventions: Drug: NNC0638-0355
- Placebo (Placebo Comparator): Participants will be randomized to receive Placebo. The study will be conducted in 4 parts. Part A: Single ascending dose (SAD). Part B,C and D: Multiple ascending dose (MAD).
  Interventions: Drug: Placebo (NNC0638-0355)

INTERVENTIONS:
Drug: NNC0638-0355 — NNC0638-0355 will be administered as a subcutaneous (s.c. under the skin) injection.
  Arms: NNC0638-0355
Drug: Placebo (NNC0638-0355) — Placebo matching NNC0638-0355 will be administered as subcutaneous (s.c. under the skin) injection.
  Arms: Placebo

SUMMARY:
The study is testing a new study medicine to treat people living with overweight or obesity. The aim of this study is to see if the medicine is safe, how it works in your body, and what your body does to the study medicine. Participants will either get the study medicine or placebo (a "dummy medicine" similar to the study medicine but without active ingredients) given as an injection under your skin. Which treatment the participants get is decided by chance. The study medicine is a potential new medicine which cannot be prescribed by doctors.

ELIGIBILITY:
Key inclusion criteria

* Male or female.
* Age 18-55 years (both inclusive) at the time of signing the informed consent.
* BMI between 25.0 and 34.9 kg/m^2 (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator.
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Key exclusion criteria

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Any condition, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* HbA1c greater than or equal to 6.5 percentage (48 mmol/mol) at screening.
* Any laboratory safety parameters at screening outside the below laboratory ranges, see designated reference range documents for specific values:

  1. Vitamin D (25-hydroxycholecalciferol) less than 12 ng/mL (30 nM) at screening
  2. Parathyroid hormone (PTH) outside normal range at screening
  3. Total calcium outside normal range at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2026-03-23 (Estimated); Study Completion 2026-09-24 (Estimated)

PRIMARY OUTCOMES:
Part A: Number of treatment emergent adverse events (TEAE) | From NNC0638-0355 administration (day 1) to completion of the end of study visit (6 weeks)
  Measured as Number of events
Part B,C,D : Number of treatment emergent adverse events (TEAE) | From first NNC0638-0355 administration (day 1) to completion of the end of study visit (20 weeks)
  Measured as Number of events

SECONDARY OUTCOMES:
Part A: AUC; area under the NNC0638-0355 plasma concentration-time curve | From NNC0638-0355 administration (day 1) to completionof the end of study visit (6 weeks)
  Measured in hours*nano mole per litre (h*nmol/L)
Part A: Cmax; maximum observed NNC0638-0355 plasma concentration | From NNC0638-0355 administration (day 1) to completionof the end of study visit (6 weeks)
  Measured in nano mole per litre (nmol/L)
Part A: t½; terminal half-life of NNC0638-0355 | From NNC0638-0355 administration (day 1) to completionof the end of study visit (6 weeks)
  Measured in hours (h)
Part B,C,D: AUC; area under the NNC0638-0355 plasma concentration-time curve | From first NNC0638-0355 administration (day 1) to completionof the end of study visit (20 weeks)
  Measured in hour*nano mole per litre (h*nmol/L)
Part B,C,D: Cmax; maximum observed NNC0638-0355 plasma concentration | From first NNC0638-0355 administration (day 1) to completionof the end of study visit (20 weeks)
  Measured in nano mole per litre (nmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- ICON, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com